CLINICAL TRIAL: NCT07120581
Title: Hyperbaric Oxygen Therapy as Salvage Therapy for Healthy, Severely Injured, Mechanically Ventilated Invasive Fungal Infection Cases Resistant to Therapy
Brief Title: Hyperbaric Oxygen Therapy Used on Severely Injured Healthy Individuals With Fungal Infections
Status: Active, not recruiting | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Reudor Grinberg, Intensive Care Physician, Assaf-Harofeh Medical Center
Other Study IDs: 0160-24-ASF
Record Dates: First submitted 2025-07-17; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Invasive Fungal Infections; Hyperbaric Oxygen Therapy
Keywords: Hyperbaric Oxygen Therapy; Invasive Fungal Infection; Trauma
MeSH Terms: conditions — Invasive Fungal Infections; Wounds and Injuries | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hyperbaric Oxygen Therapy
  Interventions: Other: Hyperbaric Oxygen Therapy

INTERVENTIONS:
Other: Hyperbaric Oxygen Therapy — Hyperbaric Oxygen Therapy at increasing pressure to 2.8 ATA for 2 hours sessions. Breaks of 5 every 20 minutes from the oxygen to air to avoid hyperoxia. Continued for the duration of the hospitalization in the ICU on a daily basis.

SUMMARY:
The goal of this observational study is to learn about the effects of Hyperbaric Oxygen Therapy on healthy individual who suffer from invasive fungal infection caused by severe trauma, who do not respond to conventional treatment. The main question it aims to answer is:

Does the treatment aid in eradicating the infection and improve the overall outcome of such patients?

ELIGIBILITY:
Inclusion Criteria:

* at least 18 year old
* Trauma as the insult type causing the infection
* Refractory IFI with failure to respond to standard therapy (medical and surgical)
* Hyperbaric Oxygen Therapy as part of the treatment

Exclusion Criteria:

* Patients who did not recieve hyperbaric oxygen therapy as part of the treatment
* Patients with immunosuppression background

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to our health care facility (Shamir Medical Center) and diagnosed with invasive fungal infection
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2024-08-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Eradication of Fungal Infectious Agent | From enrollment, baseline day 1, through study completion, an average of 4-8 weeks
  The time it takes from the start of treatments and until the first negative culture was found.

SECONDARY OUTCOMES:
Clinical Status on Discharge- ventilation status | From enrollment, baseline day 1, through study completion, an average of 4-8 weeks
  what support is the patient receiving upon discharge in terms of ventilation including invasive or non-invasive ventilation, need for oxygen or room-air
clinical status on discharge- kidney function | From enrollment, baseline day 1, through study completion, an average of 4-8 weeks
  the patient's kidney function assessed by presence of elevated Creatinine levels at discharge (mg\dl)
clinical status on discharge- Kidney function | From enrollment, baseline day 1, through study completion, an average of 4-8 weeks
  The patient's kidney function assessed by need for dialysis (yes/no)
clinical status on discharge- consciousness level | From enrollment, baseline day 1, through study completion, an average of 4-8 weeks
  evaluation of the patient's consciousness level as either alert and responsive or still requiring sedation
clinical status on discharge- wound status | From enrollment, baseline day 1, through study completion, an average of 4-8 weeks
  Whether the patient recieved a successful skin graft
clinical status on discharge- location of discharge | From enrollment, baseline day 1, through study completion, an average of 4-8 weeks
  where were the patients discharged to- regular inpatient ward, a different medical center and which department (ICU or regular inpatient), rehabilitation center or not discharged (in case of death during the hospitalization).
Adverse Events | From enrollment, baseline day 1, through study completion, an average of 4-8 weeks
  description of comlications occuring during the treatment, most notably seizures during the hyperbaric oxygen treatments

CONTACTS AND LOCATIONS:
Overall Officials: Shai Efrati, M.D, Study Director — Assaf-Harofeh Medical Center
Locations (1):
- Shamir Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arieli R, Aviner B. Acclimatization and Deacclimatization to Oxygen: Determining Exposure Limits to Avoid CNS O2 Toxicity in Active Diving. Front Physiol. 2020 Sep 4;11:1105. doi: 10.3389/fphys.2020.01105. eCollection 2020. No abstract available. PMID 33013472
- [Background] Dhingra S, Buckey JC, Cramer RA. Hyperbaric Oxygen Reduces Aspergillus fumigatus Proliferation In Vitro and Influences In Vivo Disease Outcomes. Antimicrob Agents Chemother. 2018 Feb 23;62(3):e01953-17. doi: 10.1128/AAC.01953-17. Print 2018 Mar. PMID 29229641
- [Background] Ortega MA, Fraile-Martinez O, Garcia-Montero C, Callejon-Pelaez E, Saez MA, Alvarez-Mon MA, Garcia-Honduvilla N, Monserrat J, Alvarez-Mon M, Bujan J, Canals ML. A General Overview on the Hyperbaric Oxygen Therapy: Applications, Mechanisms and Translational Opportunities. Medicina (Kaunas). 2021 Aug 24;57(9):864. doi: 10.3390/medicina57090864. PMID 34577787